CLINICAL TRIAL: NCT07388615
Title: The Effect of Echinacea (Immulant ®) in the Treatment of CRYPTOSPORIDIOSIS in Immunocompromised Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Maha Abd Elrhman, Principal Investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN000190
Record Dates: First submitted 2026-01-18; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cryptosporidium Infection
MeSH Terms: conditions — Cryptosporidiosis | interventions — Echinacea extract

STUDY DESIGN:
Intervention Model Description: open labelled randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- interventional arm (Active Comparator)
  Interventions: Drug: Echinacea Extract

INTERVENTIONS:
Drug: Echinacea Extract — Immulant ® (an extract derived from Echinacea purpurea plant)

SUMMARY:
This study aims to:

1. To evaluate the effectiveness of Immulant ® addition to standard treatment in reducing clinical symptoms of Cryptosporidiosis in immunocompromised children.
2. To measure the changes in parasite count in stool samples after treatment with Immulant ®.
3. To assess the safety and tolerability of Immulant ® in children participating in the study.

DETAILED DESCRIPTION:
The present prospective study will be (open labelled) Randomized Clinical Trial and was approved by the Research Ethical Committee Of national nutritional institute. Oral and written consent will be obtained from all patients and controls after a full explanation of the study.

A total of at least 60 immunocompromised children consecutively diagnosed with cryptosporidiosis were recruited from the outpatient clinic of National Nutritional Institute.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cryptosporidiosis Disease
* Age from 5-12 years
* Immunocompromised children
* Not receiving any drugs causing immunosuppression

Exclusion Criteria:

* Patients undergoing organ transplantation
* Patients suffering from autoimmune diseases.
* Patients suffering from hypersensitivity of this plant extract

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-18 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To measure the changes in parasite count in stool samples after treatment | six months

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutritional Institute, Cairo, Egypt